CLINICAL TRIAL: NCT05202626
Title: Detection and Biopsy Guidance of Nasopharyngeal Carcinoma Based on Artificial Intelligence and Endoscopic Images：a Multi-center Prospective Study
Brief Title: Detection and Biopsy Guidance of Nasopharyngeal Carcinoma Based on Artificial Intelligence and Endoscopic Images
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Fujian Cancer Hospital (Other Government); Hainan People's Hospital (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Chinese Academy of Sciences
Other Study IDs: CASMI002
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Nasopharyngeal Carcinoma; Image-Guided Biopsy
Keywords: Artificial Intelligence; Classification; Nasopharyngeal Carcinoma; Nasopharyngoscope; Image-Guided Biopsy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each participant exhibiting suspicious lesions during a nasopharyngeal endoscopy examination, the attending physician will determine the appropriate biopsy strategy based on the specific conditions of the lesion. The physician may opt for a single biopsy, taking a sample directly from within the lesion, or multiple biopsies, which would include one sample from inside the lesion, another from 5-8 mm outside the lesion, and a third from 8-10 mm outside the lesion. This decision will be grounded in clinical judgment and a comprehensive consideration of optimal diagnostic outcomes and patient safety.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Sun Yat-Sen University Cancer Center: The participant who is found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy in Sun Yat-Sen University Cancer Center. The physicians in Sun Yat-Sen University Cancer Center consider it necessary to perform an endoscopic image-guided biopsy.
  Interventions: Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy
- Guangdong Provincial People's Hospital: The participant who is found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy in Guangdong Provincial People's Hospital. The physicians in Guangdong Provincial People's Hospital consider it necessary to perform an endoscopic image-guided biopsy.
  Interventions: Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy
- Nanfang Hospital, Southern Medical University: The participant who is found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy in Nanfang Hospital. The physicians in Nanfang Hospital consider it necessary to perform an endoscopic image-guided biopsy.
  Interventions: Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy
- Fujian Provincial Cancer Hospital: The participant who is found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy in Fujian Provincial Cancer Hospital. The physicians in Fujian Provincial Cancer Hospital consider it necessary to perform an endoscopic image-guided biopsy.
  Interventions: Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy
- Hainan Provincial People's Hospital: The participant who is found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy in Hainan Provincial People's Hospital. The physicians in Hainan Provincial People's Hospital consider it necessary to perform an endoscopic image-guided biopsy.
  Interventions: Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal Endoscopy image-guided Biopsy — For each participant presenting with a suspicious nasopharyngeal lesion, the attending physician will assess the lesion and determine the appropriate biopsy approach. The physician may decide on multiple biopsies from the lesion area, including one sample from within the lesion itself, another from 5-8 mm outside the lesion, and a third from 8-10 mm beyond the lesion. Alternatively, a single biopsy may be deemed sufficient based on the clinical judgment. Each of these specimens will undergo pathological examination to confirm whether they are carcinomatous or non-carcinomatous.

SUMMARY:
Due to the occult anatomic location of the nasopharynx and frequent presence of adenoid hyperplasia, the positive rate for nasopharyngeal carcinoma identification during biopsy is low, thus leading to delayed or missed diagnosis for nasopharyngeal carcinoma upon initial attempt. Here, we aimed to develop an artificial intelligence tool to detect nasopharyngeal malignancies and guide biopsy under endoscopic examination based on deep learning.

DETAILED DESCRIPTION:
Due to the occult anatomic location of the nasopharynx and frequent presence of adenoid hyperplasia, the positive rate for nasopharyngeal carcinoma identification during biopsy is low, thus leading to delayed or missed diagnosis for nasopharyngeal carcinoma upon initial attempt. Here, we aimed to develop an artificial intelligence tool to detect nasopharyngeal malignancies and guide biopsy under endoscopic examination based on deep learning.

ELIGIBILITY:
Inclusion Criteria:

* The patient was found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy and the clinicans considered it necessary to perform an biopsy.
* Hemilateral lesion with limited size.

Exclusion Criteria:

* Patients with nasopharyngeal cancer, oropharyngeal cancer, hypopharyngeal cancer, etc. who have already been treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was found to have a nasopharyngeal lesion through the nasopharyngeal endoscopy and the clinican considered it necessary to perform an endoscopic image-guided biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Aera under the receiver operating characteristic curve (AUC) | three months
  AUC of an deep learning-based model in discriminating nasopharyngeal carcinoma from bengin lesion.

SECONDARY OUTCOMES:
Accuray | three months
  The agreement between the deep learning-based model and the histopathological diagnosis of the three biopsy specimens (inside the lesion, 5-8 mm outside the lesion, and 8-10 mm outside the lesion).

OTHER OUTCOMES:
Statistical significance | Three years
  Statistical significance (P value) of DFS (time from diagnosis to disease progression or death from any cause) in nasopharyngeal carcinoma patients between high-risk and low-risk group identified by deep learning-based model.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Hainan Provincial People's Hospital, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zwakenberg MA, Halmos GB, Wedman J, van der Laan BFAM, Plaat BEC. Evaluating Laryngopharyngeal Tumor Extension Using Narrow Band Imaging Versus Conventional White Light Imaging. Laryngoscope. 2021 Jul;131(7):E2222-E2231. doi: 10.1002/lary.29361. Epub 2021 Jan 4. PMID 33393666
- [Result] Li C, Jing B, Ke L, Li B, Xia W, He C, Qian C, Zhao C, Mai H, Chen M, Cao K, Mo H, Guo L, Chen Q, Tang L, Qiu W, Yu Y, Liang H, Huang X, Liu G, Li W, Wang L, Sun R, Zou X, Guo S, Huang P, Luo D, Qiu F, Wu Y, Hua Y, Liu K, Lv S, Miao J, Xiang Y, Sun Y, Guo X, Lv X. Development and validation of an endoscopic images-based deep learning model for detection with nasopharyngeal malignancies. Cancer Commun (Lond). 2018 Sep 25;38(1):59. doi: 10.1186/s40880-018-0325-9. PMID 30253801